CLINICAL TRIAL: NCT03196050
Title: Telemonitoring of Geriatric Cancer Patients Using Handheld Devices (TeleGraPH)
Brief Title: Telemonitoring of Geriatric Cancer Patients Using Handheld Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Hector-Stiftung (Other); humediQ global GmbH, Grünwald (Unknown); Vitaphone GmbH, Mannheim (Unknown)
Responsible Party: Principal Investigator, Frederik Wenz, Director and Chief Medical Officer, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TeleGraPH
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemonitoring using a handheld device (Experimental): Patients will be euqipped with either an app or a handheld device with a pre-installed app to communicate with the coordinating center.
  Interventions: Device: Handheld Device (Smart Phone)

INTERVENTIONS:
Device: Handheld Device (Smart Phone) — Handheld device will be used for 3 tasks:
  1x per day: status update ("how are you today"?)
  1x per week: 10 questions on general health status
  1x per month: EORTC QLQ-C30 questionnaire

SUMMARY:
Cancer is becoming a chronic disease, with the requirement of a lifelong intake of cancer-controlling drugs. While young(er) patients may cope with this, geriatric cancer patients may require a more customized and tailored follow up.

Most elderly patients have multiple other diseases ("comorbidities") and, due to many other factors, may per se not tolerate or simply not follow anticancer therapies. This may not only impair quality of life (QoL), but on the long rung also the therapeutic outcome (survival).

Handheld devices provide a new reporting/communication tool for patients and health care providers. TeleGraPH will assess if these devices are a suitable communication modality in a cohort of geriatric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Karnofsky Performance Status ≥ 70
* histologically confirmed malignant tumor (cancer)

Exclusion Criteria:

* concurrent severe and/or uncontrolled concomitant medical conditions
* Patients unwilling or unable to comply with using a handheld device

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Device Adherence/Compliance | 1 Year
  Frequency of using the handheld device and of daily/weekly/monthly reportings

SECONDARY OUTCOMES:
Quality of Life | 1 Year
  Assessed using the EORTC QLQ-C30 questionnaire
Reliability of reports | 1 Year
  Patient-reported status will be compared to physician-rated status

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy University Hospital Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buergy D, Siefert V, Neumaier C, Ganslandt T, Sperk E, Blessing M, Hesser J, Welzel G, Wenz F, Giordano FA. Prospective trial on telemonitoring of geriatric cancer patients using handheld devices. Strahlenther Onkol. 2020 Mar;196(3):205-212. doi: 10.1007/s00066-019-01548-0. Epub 2019 Nov 18. PMID 31740981